CLINICAL TRIAL: NCT01426646
Title: Randomized Multicenter Phase II Trial of S-1 Versus S-1 Plus Cisplatin as an Adjuvant Chemotherapy After Curative Resection of Stage II-IV(M0) Gastric Cancer
Brief Title: S-1 Versus S-1 Plus Cisplatin as an Adjuvant Chemotherapy to Treat Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Byung Woog Kang, Professor(full time instructor), Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACSPGC-01
Record Dates: First submitted 2011-01-18; First posted 2011-08-31 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; S-1; cisplatin; adjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); titanium silicide; S-1 plus cisplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S-1 treatment (Experimental): S-1 was administered at 40mg/m2 orally twice daily (days 1-28) every 42 days. Patients received a maximum of eight cycles.
  Interventions: Drug: S-1
- S-1 plus cisplatin treatment (Experimental): S-1 plus cisplatin every 3 weeks, A total of eight cycles
  * S-1: 40mg/m2 orally twice daily (days 1-14)
  * Cisplatin: 60mg/m2 IV on day 1
  Interventions: Drug: S-1 plus cisplatin

INTERVENTIONS:
Drug: S-1 — S-1 was administered at 40mg/m2 orally twice daily (days 1-28) every 42 days. Patients received a maximum of eight cycles.
  Other Names: TS-1
  Arms: S-1 treatment
Drug: S-1 plus cisplatin — S-1 plus cisplatin every 3 weeks, a total of eight cycles
  * S-1: 40mg/m2 orally twice daily (days 1-14)
  * Cisplatin: 60mg/m2 IV on day 1
  Other Names: TS-1; cisplatin
  Arms: S-1 plus cisplatin treatment

SUMMARY:
Although there has been some progress in chemotherapy for metastatic gastric cancer, no standard regimen of adjuvant chemotherapy is available, and many clinical trials have produced contradictory results. The majority of randomized clinical trials studying adjuvant chemotherapy in gastric cancer have been underpowered, involved low-volume centers, or used ineffective chemotherapy regimens. As a result, well-designed multicenter trials are still needed. The ACTS-GC trial, which demonstrated the efficacy of S-1 for stage II-III gastric cancer patients who underwent curative resection with extended lymph-node dissection (D2), may be valid in countries where D2 surgery is considered the standard of care. S-1 improved the 3-year overall survival from 70.1% for surgery alone to 80.1%. However, 3-year overall survival in stage IIIA and stage IIIB patients receiving S-1 were 77.4% and 63.4%, respectively, which are less satisfactory compared to the rate for stage II (90.7%). Based on the unsatisfactory outcome among later stage patients in the ACTS-GC adjuvant trial, further investigation is needed for more effective postoperative treatment of patients with stage IIIB and IV (M0) cancer. Therefore, the researchers investigated the efficacy and safety of S-1 versus S-1 plus cisplatin as adjuvant chemotherapy in patient with curatively resected gastric adenocarcinoma.

DETAILED DESCRIPTION:
This controlled study is designed to evaluate the efficacy of S-1 on survival compared with S-1 plus cisplatin. Patients will be randomly assigned to receive either surgery followed by treatment with S-1 plus cisplatin or surgery followed by treatment with S-1 within 42 days after curative resection. To assess the efficacy, data on recurrence and survival will be collected from the time of enrollment until 5 years after surgery. To evaluate safety, data on adverse events will be collected from the time of enrollment until 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years
2. Histologically proven adenocarcinoma of the stomach
3. Curative D2 lymphadenectomy resection for gastric cancer, who can be randomized to either study arm within 6 weeks after surgery
4. Stage II, III and IV (M0)(AJCC 7th edition)
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
6. No prior chemotherapy or radiotherapy
7. Adequate bone marrow, renal, and liver function

Exclusion Criteria:

1. Pregnant or lactating women.
2. Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-child bearing potential.
3. Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.
4. Any evidence of metastatic disease (including presence of tumor cells in the ascites).
5. Previous cytotoxic chemotherapy, radiotherapy or immunotherapy except corticosteroids, for the currently treated gastric cancer.
6. Major surgery within 4 weeks prior to study treatment start, or lack of complete recovery from the effects of major surgery.
7. History of another malignancy within the last five years except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix.

   Clinically significant (i.e. active) cardiac disease e.g. symptomatic coronary artery disease, New York Heart Association (NYHA) grade II or greater congestive heart failure or serious cardiac arrhythmia requiring medication or myocardial infarction within the last 12 months.
8. Lack of physical integrity of the upper gastrointestinal tract or those who have malabsorption syndrome likely to influence absorption of capecitabine, or inability to take oral medication.
9. Organ allografts requiring immunosuppressive therapy.
10. Serious uncontrolled intercurrent infections or other serious uncontrolled concomitant disease.
11. Prior unanticipated severe reaction to fluoropyrimidine therapy (with or without documented dihydropyrimidine dehydrogenase (DPD) deficiency) or patients with known DPD deficiency.

    Hypersensitivity to platinum compounds or any of the components of the study medications.
12. Received any investigational drug or agent/procedure, i.e. participation in another trial, within 4 weeks before randomization.
13. Blood transfusions or growth factors to aid hematologic recovery within 2 weeks prior to study treatment start.
14. Requirement for concurrent use of the antiviral agent sorivudine (antiviral) or chemically related analogues, such as brivudine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival | 3 years from enrollment.
  RFS was defined as the time from the date of surgery to relapse or death from any cause.

SECONDARY OUTCOMES:
Overall survival | 3 years from enrollment.
  OS was defined as the time from the date of surgery to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Wansik Yu, Professor, Principal Investigator — Kyungpook National University Hospital
Locations (2):
- South Korea (2):
  - Donga university hospital, Busan
  - Ulsan University Hospital, Ulsan